CLINICAL TRIAL: NCT02481180
Title: An Open, Dose Escalation, Multiple Dose Study to Assess Tolerance、Pharmacokinetics、Preliminary Efficacy of T0001 in RA (Rheumatoid Arthritis)
Brief Title: Tolerance, Pharmacokinetics and Preliminary Efficacy of T0001 in RA (Rheumatoid Arthritis)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T0001-P2.0
Record Dates: First submitted 2015-06-18; First posted 2015-06-25 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — T0001; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T0001 (Experimental)
  Interventions: Drug: T0001
- Enbrel (Active Comparator)
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: T0001 — injection (SC) T0001 15mg weekly for 12 weeks
  Arms: T0001
Drug: T0001 — injection (SC) T0001 30mg weekly for 12 weeks
  Arms: T0001
Drug: T0001 — injection (SC) T0001 30mg every two weeks for 12 weeks
  Arms: T0001
Drug: T0001 — injection (SC) T0001 50mg every two weeks for 12 weeks
  Arms: T0001
Drug: Enbrel — injection (SC) enbrel 50mg twice a week for 12 weeks
  Arms: Enbrel

SUMMARY:
The purpose of this study is to assess the MTD, Pharmacokinetics and preliminary efficacy of T0001 in Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years old;
* Diagnosed with active RA;
* DMARDs therapy must not be used for at least 28 days prior to baseline;
* If a patient has received NSAIDs，current NSAIDs therapy must have been at a stable dose for at least 28 days prior to baseline;
* Patient or patient's legal representative able to give written informed consent for participation in the trial.

Exclusion Criteria:

* Acute or chronic infection, or history of active tuberculosis;
* History of diseases of central nervous system, cardiovascular system, kidney, liver ( specified liver function index), digestive system, respiratory system , metabolism system;
* Patients who have a high risk of infection (with a current infectious disease, a chronic infectious disease, a history of serious infectious disease);
* Patients who use 5 Unit doses tuberculin skin test are positive( 48-72 hour scleroma reading≥5mm);
* Patients who currently have, or who have a history of, malignancy;
* Patients who lack of understanding ,communication or collaboration, and can't comply with the protocols;
* Female patients who are breastfeeding or pregnant, who are of childbearing potential.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerance Dose | 4 weeks
Peak Plasma Concentration (Cmax) | 14 weeks
Area under the plasma concentration versus time curve (AUC) | 14 weeks
steady-state concentration（Css） | 14 weeks

SECONDARY OUTCOMES:
American College of Rheumatology 20% (ACR20) Response | 12 weeks
  ACR20 responders are subjects with at least 20% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1)Health Assessment Questionnaire-Disability Index (HAQ-DI), 2)C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS)
American College of Rheumatology 50% (ACR50) Response | 12 weeks
  ACR50 responders are subjects with at least 50% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1)Health Assessment Questionnaire-Disability Index (HAQ-DI), 2)C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS)
American College of Rheumatology 70% (ACR70) Response | 12 weeks
  ACR70 responders are subjects with at least 70% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1)Health Assessment Questionnaire-Disability Index (HAQ-DI), 2)C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Li zhan Guo, Ph.D, Principal Investigator — Peking University People's Hospital; wang wei, Study Director — Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd.
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Shen Y, Li G, Gu C, Chen B, Chen A, Li H, Gao B, Liang C, Wu J, Yang T, Jin L, Su Y. T0001, a variant of TNFR2-Fc fusion protein, exhibits improved Fc effector functions through increased binding to membrane-bound TNFalpha. PLoS One. 2017 May 19;12(5):e0177891. doi: 10.1371/journal.pone.0177891. eCollection 2017. PMID 28542350